CLINICAL TRIAL: NCT06288204
Title: Association of Green Propolis Extract and Royal Jelly to Modulate Inflammation and Oxidative Stress in Hypertensive Patients and/or With Chronic Kidney Disease
Brief Title: Green Propolis Extract and Royal Jelly in Hypertensive Patients and/or With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Denise Mafra16
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases; Hypertension; Cardiovascular Diseases
Keywords: chronic kidney disease; hypertension; cardiovascular disease; inflammation; oxidative stress; green propolis; royal jelly; Nrf2; Nuclear factor kappa-B
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Cardiovascular Diseases; Inflammation | interventions — royal jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propolis associated with Royal Jelly Group (Experimental): 4 capsules a day, providing daily royal jelly in an amount of 100 mg/day plus 500 mg/day of propolis together, for 2 months.
  Interventions: Dietary Supplement: Propolis associated with Royal Jelly
- Royal Jelly (Experimental): Royal Jelly will receive 1 capsule a day, providing daily royal jelly in an amount of 100 mg/day, for 2 months.
  Interventions: Dietary Supplement: Royal Jelly
- Placebo (Placebo Comparator): 4 capsules a day of placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Propolis associated with Royal Jelly — The participants will consume 4 capsules a day, providing daily royal jelly in an amount of 100 mg/day plus 500 mg/day of propolis together, for 2 months.
  Arms: Propolis associated with Royal Jelly Group
Dietary Supplement: Royal Jelly — The participants will consume 1 capsules a day, providing daily royal jelly in an amount of 100 mg/day, for 2 months.
  Arms: Royal Jelly
Dietary Supplement: Placebo — The participant will consume 4 capsules a day of placebo, for 2 months.
  Arms: Placebo

SUMMARY:
This work aims to evaluate the effects of the association of green propolis extract with royal jelly on inflammation and oxidative stress in participants with chronic kidney diseases (CKD) and Systemic arterial hypertension (SAH), in a longitudinal, randomized, double-blind, placebo-controlled clinical trial that will be carried out for 2 months.

DETAILED DESCRIPTION:
Propolis and royal jelly are bee products. Propolis is a resinous mixture produced by bees with their saliva and the addition of wax, from exudates collected from buds and plant sap. Royal jelly is a substance produced in the hypopharyngeal glands of young worker bees. Both products are rich in bioactive compounds such as polyphenols. The combination of propolis extract and royal jelly, substances constituted by the combination of several chemical components with potential biological activity, may emerge as a promising adjuvant therapeutic alternative for patients with CKD and SAH.

ELIGIBILITY:
Inclusion Criteria:

* patients in stages 3 and 5 of CKD (GFR from 15 to 59 mL/min),
* patients receiving ambulatorial nutrition treatment at least 6 months
* patients on regular Hemodialysis treatment for at least 6 months
* patients using one to three antihypertensive drugs

Exclusion Criteria:

* autoimmune and infectious diseases,
* diabetes
* cancer
* AIDS
* pregnant women
* patients using catabolic drugs or antibiotics;
* patients with catheter access to hemodialysis;
* patients using antioxidant vitamin supplements, prebiotics, probiotics, symbiotic,
* Patients on regular intake of propolis who are allergic to corn starch or report being allergic to bee stings.
* patients with acute myocardial infarction (AMI) and/or cerebrovascular accident (CVA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in factor nuclear kappaB | Baseline and 8 weeks (2 months)
  Get blood samples to evaluate the supplementation effects in factor nuclear kappaB by quantitative real-time polymerase chain reaction.
Change in intestinal microbiota | Baseline and 8 weeks (2 months)
  Stool samples will be collected to evaluate the taxa of bacteria colonizing the intestinal microbiota through short-read sequencing of the V4 region of the RNA ribosomal (rRNA) gene on the Illumina platform.

SECONDARY OUTCOMES:
Change in senescence biomarkers | Baseline and 8 weeks (2 months)
  Get blood samples to evaluate the supplementation effects in p14, p16, p21, p53.
Change in uremic toxins | Baseline and 8 weeks (2 months)
  Get blood samples to evaluate the supplementation effects in p-cresyl sulfate (p-CS)

OTHER OUTCOMES:
Change in adhesion molecules | Baseline and 8 weeks (2 months)
  Get blood samples to evaluate the supplementation effects Vascular Cell Adhesion Molecule (VCAM).
Change in blood pressure | Baseline and 8 weeks (2 months)
  Evaluate at baseline and 8 weeks the Systolic or Diastolic Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Participant data will not be public to other research unless necessary.